CLINICAL TRIAL: NCT00984802
Title: A Prospective, Randomized, Comparative, Blinded, Placebo-Controlled, Three Different Intravenous Dose, Phase 2a Study of the Safety and Efficacy of CMX-2043 in Subjects Undergoing PCI and Peri-Operative Reperfusion Treatment (SUPPORT-1)
Brief Title: Safety and Efficacy of CMX-2043 in Subjects Undergoing Coronary Reperfusion Therapy
Acronym: SUPPORT-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ischemix, LLC (Industry)
Responsible Party: Duffy Dufresne, Ischemix, LLC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMX-2043-2a
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Stable Coronary Artery Disease; Percutaneous Coronary Intervention
MeSH Terms: interventions — alpha-N-(1,2-dithiolane-3-pentanoyl)glutamylalanine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low dose (Experimental)
  Interventions: Drug: CMX-2043
- Mid Dose (Experimental)
  Interventions: Drug: CMX-2043
- High Dose (Experimental)
  Interventions: Drug: CMX-2043
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: CMX-2043 — Solution for IV administration at 0.8, 1.6 or 2.4 mg/kg single dose.
  Arms: High Dose; Low dose; Mid Dose
Drug: Placebo control — Vehicle solution for IV administration single dose.
  Arms: Placebo

SUMMARY:
This study is conducted to assess the safety of CMX-2043 solution for intravenous (IV) injection, and to evaluate efficacy on the basis of the changes seen in the cardiac biomarkers and continuous electrocardiography (ECG) monitoring. Additionally, correlation of the levels/changes in the biomarkers and the pharmacokinetic evaluations of the drug will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have stable coronary artery disease undergoing elective PCI.
* Female subjects not of child-bearing potential.
* Absence of ST segment depression >1.0 mm and absence of ST elevation >1.0 mm in any lead on the baseline 12-lead ECG.
* subjects with CK-MB and troponin-T levels lower than the upper limit of normal.
* Subjects free of acute injuries or illnesses.

Exclusion Criteria:

* Subjects with unstable angina (angina at rest, worsening frequency, duration of angina) or other signs of unstable coronary artery disease.
* Subjects who had had an MI within 14 days prior to the PCI procedure.
* Subjects with conditions that contraindicate the PCI (e.g. coagulopathy, valvular disease, PVD).
* Subjects with history of TIA/stroke within 90 days or any intracranial bleed.
* Subjects with creatinine clearance ≥ 1.5 times the upper limit of normal.
* Subjects with an active history of psychiatric disorders that is likely to limit the validity of consent to participate in the study or limit the ability to comply with the protocol requirements.
* Subjects with a history of alcohol or drug abuse.
* Subjects with documented history of human immunodeficiency virus (HIV), or Hepatitis B (HBsAg) or Hepatitis C (HCV) virus positive.
* Subjects with uncorrected clinically significant abnormalities of clinical laboratory tests who in the investigators opinion will interfere with the study conduct.
* Subject with chronic diseases considered by the anesthetist unfit for surgery and/or who in the opinion of the investigator will increase the risk of the study or obscure the interpretation of results.
* Subjects who have participated in a clinical study within 1 month or are currently participating in a clinical study of an investigational agent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Safety as measured by changes in CK-MB | within 24 hours

SECONDARY OUTCOMES:
Cardiac biomarkers | within 24 hours
ST segment changes | within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alan S. Lader, Ph.D., Study Director — Ischemix, LLC
Locations (5):
- United States (2):
  - St. Vincent Hospital, Worcester, Massachusetts
  - Duke University Hospital, Durham, North Carolina
- India (3):
  - Madras Medical Mission, Chennai
  - Hinduja Hospital, Mumbai
  - Poona Hospital, Pune